CLINICAL TRIAL: NCT05793281
Title: A Retrospective Observational Study to Investigate the Prevalence of NTRK Gene Fusion Positive in Solid Tumor in Japan
Brief Title: An Observational Study to Learn More About NTRK Gene Fusion Positive in Solid Tumor in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22415
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Advanced or Recurrent Solid Tumor Harboring an NTRK Gene Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with solid tumor and genome profiling results: Retrospective data analysis, the dataset for this study will be extracted from the C-CAT database.
  Interventions: Other: No Drug

INTERVENTIONS:
Other: No Drug — Retrospective data analysis, the dataset for this study will be extracted from the C-CAT database.

SUMMARY:
This is an observational study in which data from the past of people with solid tumors harboring an NTRK gene fusion in Japan are studied. In observational studies, only observations are made without specified advice or interventions.

Advanced or recurrent solid tumor harboring an NTRK gene fusion is a rare type of solid cancer caused by specific changes in the genes called NTRK gene fusion, and which has spread to nearby tissues and/or lymph nodes or has returned. Due to this change in the gene, an altered protein known as a TRK fusion protein is made, which can cause cancer cells to grow and survive.

The main purpose of this study is to learn more about NTRK gene fusion in people in Japan. To do this, researchers will collect information on the number or percentage of Japanese people with NTRK gene fusion in any solid tumor.

The data will come from the national database called C-CAT. They will cover the period from June 2019 until January 2023.

Besides this data collection, no further tests or examinations are planned, and no visits are required in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any solid tumor and genome profiling results

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with any solid tumor and genome profiling results
Sampling Method: Non-Probability Sample
Enrollment: 46621 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of patients with NTRK gene fusions by patient characteristic categories, such as tumor types | Retrospective data analysis from June 2019 to the latest data available (planned end of February 2023)
Distribution of cancer types in patients with NTRK fusion positive among all, adult and pediatric | Retrospective data analysis from June 2019 to the latest data available (planned end of February 2023)

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.